CLINICAL TRIAL: NCT06719999
Title: Box for Health by Tradition & Innovation (B4HT): Promoting Sustainable Mediterranean Diet by Healthy Foods
Brief Title: PRIMA Project- Box for Heath and Tradition (B4HT)
Acronym: PRIMA-B4HT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, piero portincasa, Full Professor, University of Bari
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRIMA2023
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Obesity and Obesity-related Medical Conditions
Keywords: Mediterranean lunch boxes; Obesity; Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Lean, ongoing diet (n=40) (No Intervention)
- Lean, B4HT (n= 40) (Experimental): B4HT Mediterranean Lunch box
  Interventions: Dietary Supplement: B4HT Mediterranean Lunch box
- OW/OB without prediabetes/T2DM ongoing diet (n=40) (No Intervention)
- OW/OB without prediabetes/T2DM, B4HT (n= 40) (Experimental): B4HT Mediterranean Lunch box
  Interventions: Dietary Supplement: B4HT Mediterranean Lunch box
- OW/OB, with prediabetes/T2DM, ongoing diet (n=40) (No Intervention)
- OW/OB with prediabetes/T2DM, B4HT (n= 40) (Experimental): B4HT Mediterranean Lunch box
  Interventions: Dietary Supplement: B4HT Mediterranean Lunch box

INTERVENTIONS:
Dietary Supplement: B4HT Mediterranean Lunch box — lunch boxes developed in the PRIMA project (L-MedFood or F-MedFood, ~600 kcal)
  Arms: Lean, B4HT (n= 40); OW/OB with prediabetes/T2DM, B4HT (n= 40); OW/OB without prediabetes/T2DM, B4HT (n= 40)

SUMMARY:
The study aims to explore the effects of a tailored nutritional intervention for maintaining (normal-weight subjects) or reducing (overweight or obese subjects) body weight. In a subgroup of patients with prediabetes/T2DM, the effect of the nutritional intervention by Mediterranean lunch boxes developed in the PRIMA project on gluco-lipid homeostasis will be also evaluated. Secondary objectives are to evaluate the nutritional and functional benefits of the intervention strategies on pathogenetic factors affecting metabolic and pro-inflammatory status and intestinal permeability.

DETAILED DESCRIPTION:
Protocol summary The study aims to explore the effects of a tailored nutritional intervention for maintaining (normal-weight subjects) or reducing (overweight or obese subjects) body weight. In a subgroup of patients with prediabetes/T2DM, the effect of the nutritional intervention by Mediterranean lunch boxes developed in the PRIMA project on gluco-lipid homeostasis will be also evaluated. Secondary objectives are to evaluate the nutritional and functional benefits of the intervention strategies on pathogenetic factors affecting metabolic and pro-inflammatory status and intestinal permeability.

Patients All enrolled participants (n=450, age 25-65) will undergo, following written informed consent, a 12-weeks, controlled, randomized, multicenter clinical study with multiple arms conducted on normal weight, overweight or obese subjects with or without prediabetes or other metabolic risk factors in Italy and Lebanon.

Study design Participants will be assigned to the healthy group (HG, n= 150) or to the dysmetabolic group (DG, n=300) according to a previous clinical assessment. The two groups will be comparable for age/gender composition. In each group, subjects will be randomized to continue the ongoing diet (controls) or to receive one of the lunch boxes developed in the project (L-MedFood or F-MedFood, ~600 kcal) 3-times/week during 12 weeks (treatment). In the treated groups, healthy subjects will receive the L-MedFood lunch box, the overweight/obese subjects, with or without prediabetes/T2DM, will receive the F-MedFood Box. The consumption of lunch boxes will be associated, in all enrolled subjects, with the use of iMFood, an interactive and easy-to-understand APP developed in this project and fulfilling the goal of a new Agro-Food Value Chain solution, to enable the transition to healthy and sustainable dietary behavior.

Groups

The different arms of the study will be as follows:

* Group 1: Lean, ongoing diet (n=40);
* Group 2: Lean, B4HT (n= 40);
* Group 3: OW/OB without prediabetes/T2DM ongoing diet (n=40);
* Group 4: OW/OB without prediabetes/T2DM, B4HT (n= 40);
* Group 5: OW/OB, with prediabetes/T2DM, ongoing diet (n=40);
* Group 6: OW/OB with prediabetes/T2DM, B4HT (n= 40). Participants will have follow-up phone/physical visits every third week (4 visits). These subjects will receive Fat-Dysmetabolic Box (3-times/week) and APP iMFood with standard-of-care pharmacological treatments.

Duration The study is planned to last 12 weeks.

Outputs In all arms of the study, the primary outcomes are weight loss and satisfaction index. Secondary outcomes include changes in gluco-lipid homeostasis and in visceral and liver fat quantitative ultrasonography, adherence to Mediterranean diet (assessed and monitored by the validated score MEDI-LITE). Exploratory analyses will include analyses of inflammatory status, intestinal permeability as assessed by oral quadruple test ingestion, gut microbiota profile and metabolomic analysis. Cause-and-effect relationships between B4HT and risk reduction and decrease in obesity rate and other metabolic abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Subjects able to provide Informed Consent
* Age over 18 years

Exclusion Criteria:

* Lack of informed consent
* Pregnancy
* Chemotherapy
* Participation in other research protocols.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Weight (Kg) | From enrollment to the end of treatment at 12 weeks
  The primary outcome isweight loss

SECONDARY OUTCOMES:
Fasting glucose | From enrollment to the end of treatment at 12 weeks
  Change in glycemic profile
Lipid profile (TC, TG, LDL, HDL) | From enrollment to the end of treatment at 12 weeks
  Change in Lipid profile
Liver enzymes | From enrollment to the end of treatment at 12 weeks
  Change in AST, ALT, and GGT
Abdominal fat storage | From enrollment to the end of treatment at 12 weeks
  Change in abdominal fat depostion
Liver steatosis | From enrollment to the end of treatment at 12 weeks
  Assesment of liver fat accumulation

OTHER OUTCOMES:
Inflammatory markers | At baseline and at the end of treatment (12 weeks)
  Assessment of serum inflammatory markers such as Interleukins and cytokines
Gut Microbiota | At baseline and at the end of treatment (12 weeks)
  Assessment of fecal gut microbiota composition

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico di Bari, Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Portincasa P, Khalil M, Mahdi L, Perniola V, Idone V, Graziani A, Baffy G, Di Ciaula A. Metabolic Dysfunction-Associated Steatotic Liver Disease: From Pathogenesis to Current Therapeutic Options. Int J Mol Sci. 2024 May 22;25(11):5640. doi: 10.3390/ijms25115640. PMID 38891828
- [Background] Santoro S, Khalil M, Abdallah H, Farella I, Noto A, Dipalo GM, Villani P, Bonfrate L, Di Ciaula A, Portincasa P. Early and accurate diagnosis of steatotic liver by artificial intelligence (AI)-supported ultrasonography. Eur J Intern Med. 2024 Jul;125:57-66. doi: 10.1016/j.ejim.2024.03.004. Epub 2024 Mar 14. PMID 38490931
- [Background] Abdallah H, Khalil M, Farella I, JohnBritto JS, Lanza E, Santoro S, Garruti G, Portincasa P, Di Ciaula A, Bonfrate L. Ramadan intermittent fasting reduces visceral fat and improves gastrointestinal motility. Eur J Clin Invest. 2023 Sep;53(9):e14029. doi: 10.1111/eci.14029. Epub 2023 May 19. PMID 37203871
- [Background] Khalil M, Abdallah H, Razuka-Ebela D, Calasso M, De Angelis M, Portincasa P. The Impact of Za'atar Antioxidant Compounds on the Gut Microbiota and Gastrointestinal Disorders: Insights for Future Clinical Applications. Antioxidants (Basel). 2023 Feb 9;12(2):426. doi: 10.3390/antiox12020426. PMID 36829984
- [Background] Khalil M, Shanmugam H, Abdallah H, John Britto JS, Galerati I, Gomez-Ambrosi J, Fruhbeck G, Portincasa P. The Potential of the Mediterranean Diet to Improve Mitochondrial Function in Experimental Models of Obesity and Metabolic Syndrome. Nutrients. 2022 Jul 28;14(15):3112. doi: 10.3390/nu14153112. PMID 35956289
- [Background] Portincasa P, Bonfrate L, Khalil M, Angelis M, Calabrese FM, D'Amato M, Wang DQ, Di Ciaula A. Intestinal Barrier and Permeability in Health, Obesity and NAFLD. Biomedicines. 2021 Dec 31;10(1):83. doi: 10.3390/biomedicines10010083. PMID 35052763